CLINICAL TRIAL: NCT03928392
Title: Does an Occupational Therapy Program Enhance Mental Health Outcomes for Veterans Who Scuba Dive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5180305
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Post Traumatic Stress Disorder; Depression; Anxiety; Stress, Psychological
Keywords: Post Traumatic Stress Disorder, Depression, Anxiety, Stress, SCUBA, Occupational therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Stress, Psychological | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: There are two groups for this study. Both groups will engage in two SCUBA dives. Additionally one group will receive occupational therapy and the other will not. The occupational therapy sessions will occur in conjunction with the SCUBA dive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCUBA Dive with OT (Experimental): Two SCUBA dives in conjunction with occupational therapy intervention. The occupational therapy intervention will take place on the beach or on the boat before/after the SCUBA dive. The intervention will consist of learning 3 different breathing techniques. Participants will also be educated about mindfulness principals. Additionally, participants will complete journaling activities between dives.
  Interventions: Behavioral: SCUBA with Occupational Therapy (OT)
- SCUBA Dive without OT (Active Comparator): The group will engage in two SCUBA dives.
  Interventions: Behavioral: Self-Contained Underwater Breathing Apparatus (SCUBA) without OT

INTERVENTIONS:
Behavioral: SCUBA with Occupational Therapy (OT) — Study participants will complete two OT sessions in conjunction to their regular SCUBA diving activity. OT intervention includes breathing techniques, mindfulness strategies and a journal activity.
  Arms: SCUBA Dive with OT
Behavioral: Self-Contained Underwater Breathing Apparatus (SCUBA) without OT — Study participants will continue their regular SCUBA diving activity through the Wounded American Veterans Experience SCUBA (WAVES) program. They will complete two dives.
  Arms: SCUBA Dive without OT

SUMMARY:
The purpose of the study is to investigate whether an occupational therapy program could enhance mental health outcomes for veterans who SCUBA dive. SCUBA diving requires modified breathing techniques and has been found to provide calming effects to individuals who engage in this activity. Occupational therapy interventions such as mindfulness, journaling, and deep breathing techniques can also provide similar calming effects. Therefore, this study will explore whether occupational therapy can provide additional benefits to overall mental health of veterans who SCUBA dive.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 95 years of age
* Participation in WAVES Project for at least 3 months
* Completion of 3 open water dives
* Proficient in written and verbal English

Exclusion Criteria:

* Younger than 18 years of age or older than 95 years of age
* Not a member of WAVES Project within 3 months of study recruitment
* Has not completed 3 open water dives
* Not proficient in written and verbal English

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Krpalek, PhD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCUBA Dive With OT | SCUBA Dive Without OT
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCUBA Dive With OT | SCUBA Dive Without OT | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.29 (7.97) | 40.63 (7.67) | 42.33 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Occupational Performance
Description: Study participants will complete the assessment, Canadian Occupational Performance Measure (COPM) which is an individualized composite measurement of factors designed to assess clients' perception of their occupational performance and satisfaction with that performance. The participants will identify up to 5 goals. For each goal the participant will rate their perceived performance on a scale of 1 to 10, with 1 representing the lowest level of performance and 10 representing the highest level of performance. The average of the scores will be recorded. Participants will also rate their satisfaction with performance on a scale of 1 to 10, with 1 representing the lowest level of satisfaction and 10 representing the highest level of satisfaction. The average of these scores will represent the satisfaction with performance score.
Time Frame: Change between baseline and three weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCUBA Dive With OT | SCUBA Dive Without OT
Number analyzed (Participants) | 7 | 8
score on a scale | 4.2 (.4) | 4.1 (.4)

2. Secondary Outcome: The PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) assesses the 20 DSM-5 symptoms of PTSD through a 20-item self-report measure. In the PCL-5, individuals are presented with a list of problems people may have as a result of a stressful situation. Individuals are asked to indicate how much they have been bothered by this problem in the past month. Problems can be rated as "not at all, a little bit (1), moderately (2), quite a bit (3), or extremely" (4). A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Higher scores reflect more PTSD symptoms. Initial research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD across samples.
Time Frame: Change between baseline and three weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCUBA Dive With OT | SCUBA Dive Without OT
Number analyzed (Participants) | 7 | 8
score on a scale | 21.6 (7.3) | 30.3 (6.8)

3. Secondary Outcome: The Depression Anxiety and Stress Scales (DASS)
Description: The Depression Anxiety and Stress Scales (DASS) is a individualized composite measurement used to assess symptoms of depression, anxiety, and stress in community settings. The DASS-21 asks 21 questions and is comprised of three subscales: The Depression sub-scale which measures hopelessness, low self-esteem, and low positive affect; the Anxiety scale which assesses autonomic arousal, musculoskeletal symptoms, situational anxiety and subjective experience of anxious arousal; and the Stress scale which assesses tension, agitation, and negative affect. There are 21 questions and responses are provided on a 4-point Likert scale, Where 0 = Did not apply to me, 1 = applied to me some degree, or some of the time, 2 = applied to me a considerable degree or good part of time, and 3 = applied to me very much or most of the time. The three subscales can be totaled for an overall DASS score, ranging from 0 to 63, with higher scores indicating higher levels of symptoms.
Time Frame: Change between baseline and three weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCUBA Dive With OT | SCUBA Dive Without OT
Number analyzed (Participants) | 7 | 8
score on a scale | 28.00 (32.86) | 36.12 (25.22)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | SCUBA Dive With OT | SCUBA Dive Without OT
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03928392/Prot_SAP_000.pdf